CLINICAL TRIAL: NCT00888199
Title: Clinical Trial of Tensegrity Prosthetics K3 Promoter Foot Prosthesis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tensegrity Prosthetics (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Jerome Rifkin/CEO & CTO, Tensegrity Prosthetics
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1-Rifkin
Record Dates: First submitted 2009-04-23; First posted 2009-04-27 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Amputation
Keywords: amputation; amputee; prosthetic; foot; prosthesis; Tensegrity; Prosthetics; K3 Promoter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Congenital/Traumatic (Experimental): Individuals who were born with a limb deficiency or who have had a traumatic amputation.
  Interventions: Device: Experimental prosthetic foot (K3 Promoter)
- Dysvascular/Diabetic (Experimental): Individuals who have had an amputation as a result of vascular disease.
  Interventions: Device: Experimental prosthetic foot (K3 Promoter)

INTERVENTIONS:
Device: Experimental prosthetic foot (K3 Promoter) — Experimental prosthetic foot

SUMMARY:
The purpose of this clinical trial is to determine if the experimental Tensegrity prosthetic foot offers a reduction of the amount of oxygen used while walking, if stability is improved over current prosthetic feet, and whether the experimental device actually increases activity in amputees.

DETAILED DESCRIPTION:
Tensegrity Prosthetics' objectives are to test whether the K3 Promoter prosthetic foot affects walking efficiency or stability in trans-tibial unilateral amputees when compared to their current prostheses. The primary objectives are to determine if the experimental foot changes Cost of Transport (ml O2/kg/meter) or Stride Time Variability compared to an amputee's current prosthesis. Cost of Transport is an indicator of metabolic efficiency and Stride Time Variability indicates how likely a person is to fall. Oxygen consumption and stride time will be collected on a treadmill at the Gait and Motion Lab at the University of Colorado in Boulder.

ELIGIBILITY:
Inclusion Criteria:

1. K2 or K3 classification based on current prosthetic device.
2. Males and females ≥ 18 years of age
3. Willing and able to sign informed consent
4. Able to read, write, and speak English
5. Documented to have a unilateral trans-tibial amputation
6. Actively utilizing a definitive prosthesis for at least 12 months
7. Utilizing current prosthetic foot for at least 3 months
8. Cognitively functional, in the opinion of the prosthetists'
9. Able to maintain a good gait on their existing limb for approximately 45 minutes
10. have a healthy residual limb in good condition
11. have a socket with a good, trouble-free fit on their residual limb

Exclusion Criteria:

1. Significant ulcers or infections associated with a compromised circulation of the other lower limb
2. Intermittent Claudication or Critical Leg Ischemia in the non-amputated leg
3. K0, K1or K4 Classification
4. Irreducible, pronounced knee or hip flexion contractures
5. Bilateral amputations
6. Use of a walker for ambulation
7. Severe arthritis that would limit the ability to stand without pain or discomfort or the subject's ability to ambulate is limited by symptoms other than the prothesis (e.g., shortness of breath, fatigue, angina, arthritis, etc.). If, in the opinion of the investigator, the subject were to improve their ability to ambulate from the K3 Promoter to the extent that his or her walking would then be limited by a symptom other than the prothesis, the subject should not be enrolled
8. Any other clinically significant medical or psychiatric condition that in the opinion of the Investigator could impact the subject's ability to successfully complete this trial
9. Advanced neurologic disorder
10. Severe congestive heart failure, angina pectoris, or obstructive pulmonary disease
11. Use of medication that causes impaired balance or judgment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Change in metabolic cost of transport | 30 and 60 days after the beginning of the protocol
Stride time variability | 30 and 60 days after beginning of protocol

SECONDARY OUTCOMES:
Amputee Mobility Predictor Questionnaire | Beginning and end of protocol
Actual change in activity as measured by a step counter | throughout protocol (60 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Rifkin, MS ME, Principal Investigator — Tensegrity Prosthetics
Locations (1):
- University of Colorado Gait Lab, Boulder, Colorado, United States